CLINICAL TRIAL: NCT00519493
Title: A Two Part Study: An Investigator-initiated, Single-center, Single-blinded, Randomized Clinical Study Comparing Two Closure Techniques of Excised Keloids
Brief Title: A Randomized Clinical Study Comparing Two Closure Techniques of Excised Keloids
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Issues with application of Clozex intervention
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Robert S. Kirsner, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20061027
Record Dates: First submitted 2007-08-21; First posted 2007-08-22 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Keloid
Keywords: Clozex; Sutures
MeSH Terms: conditions — Keloid | interventions — Sutures

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suture (Active Comparator): A keloid will be surgically excised and the surgical wound generated will be randomized to be closed with sutures.
  Interventions: Procedure: Suture
- Clozex (Active Comparator): One keloid will be surgically excised and the surgical wound generated will be randomized to be closed with Clozex.
  Interventions: Device: Clozex

INTERVENTIONS:
Procedure: Suture — One keloid will be surgically excised and the surgical wound generated will be randomized to be closed with sutures.
  Arms: Suture
Device: Clozex — One keloid will be surgically excised and the surgical wound generated will be randomized to be closed with Clozex.
  Arms: Clozex

SUMMARY:
This investigator initiated study, single-blinded, parallel, randomized study will be conducted in subjects with 2 or more keloids similar in size and duration on a similar area of the body. The response of the closure techniques will be evaluated by clinical and instrumental assessments. Each qualified subject will be assessed and the keloids will be randomly assigned to the Clozex or suture closure. One keloid will be surgically excised and the surgical wound generated will be randomized to be closed with Clozex. A second keloid will be surgically excised and the surgical wound generated will be randomized to be closed with sutures. The inflammation index and the keloid recurrence rate at each surgical wound closure site will be compared.

DETAILED DESCRIPTION:
This study will be undertaken to compare the efficacy of two closure techniques for excised keloids. (1) Clozex, a non-latex, hypoallergenic adhesive polymeric interlaced film designed to adhere to proximal wound edges for 7-10 days, will be used after the punch biopsy or excision of a keloid and (2) sutures to close a similar second keloid after the punch biopsy or excision of a keloid.

On day 12, the investigator and subject will assess the keloid site(s) with the use of a visual analog scale.

There is an optional follow-up at 3 months and 6 months to assess the recurrence of the keloid and the effectiveness of the treatments with a visual analog scale.

The subject will assess the keloid site(s) with the use of the following visual analog scale:

1. Cosmetic appearance
2. Pain
3. Tenderness
4. Itching
5. Oozing
6. Redness
7. Warmth

The investigator will assess the keloid site(s) with the use of this visual analog scale:

1. Global appearance
2. Color
3. Matte/Shiny
4. Contour
5. Distortion
6. Texture
7. Oozing
8. Redness
9. Warmth
10. Firmness

ELIGIBILITY:
Inclusion Criteria:

* Male or females, in good health, and at least 12 years of age.
* Individuals with 2 or more keloids on the trunk, arm, leg, and neck between 0.5 and 2 cm in length.
* Individuals who are willing and able to participate in the requirements of the study, including signing the informed consent.
* In the opinion of the investigator, the 2 keloids can be excised in a similar manner and closed properly with the two techniques and will benefit from the procedure.
* In the opinion of the investigator, the keloid could benefit from surgical procedure.

Exclusion Criteria:

* Individuals with keloids that do not fit into the criteria.
* Individuals who are planning pregnancy, pregnant, or breast feeding.
* Individuals with a history of medical or dermatologic conditions which, in the opinion of the investigator, would put the subject at heightened risk or would limit complicate the study evaluations required by the protocol.
* Individuals who present with excessive body hair in the designed keloid area.
* Individuals with uncontrolled diabetes.
* Individuals with autoimmune disorders (HIV/AIDs, SLE).
* Subjects who have received keloid treatment within one month of the first day of the study.
* Individuals who plan to receive keloid treatment(s) during the study.
* Individuals who are currently taking prescription or over the counter medication or interventions on a regular basis that as part of their mechanism of action, have the potential to mask an inflammatory reaction. Examples of such medications include, but are not limited to, corticosteroids, non-steroid anti-inflammatory drugs (NSAIDs), antihistamines, aspirin (81mg or less daily dosage permissible), or other medications that in the opinion of the investigator or designee may expose the subject to heightened risk or complicate the study assessments.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Global appearance at Keloid site. | 12 (+/-2) days after excision of keloid

SECONDARY OUTCOMES:
Global appearance at Keloid site. | 3 months (+/-3 weeks)
Global appearance at Keloid site. | 6 months (+/-4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Berman, M.D., Ph.D., Principal Investigator — University of Miami Department of Dermatology and Cutaneous Surgery
Locations (1):
- Skin Research Group Office, Miami, Florida, United States

REFERENCES:
- [Background] Beausang E, Floyd H, Dunn KW, Orton CI, Ferguson MW. A new quantitative scale for clinical scar assessment. Plast Reconstr Surg. 1998 Nov;102(6):1954-61. doi: 10.1097/00006534-199811000-00022. PMID 9810991
- See also: Homepage of Skin Research Group — http://www.skininvestigation.com